CLINICAL TRIAL: NCT05099380
Title: Validation of Senofilcon A With New UV / HEV Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6470
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST lens (Experimental): Eligible subjects that are habitual wearers of silicone hydrogel spherical contact lenses will be randomized to the TEST Lens for the duration of the study.
  Interventions: Device: senofilcon A C3
- CONTROL lens (Active Comparator): Eligible subjects that are habitual wearers of silicone hydrogel spherical contact lenses will be randomized to the CONTROL Lens for the duration of the study.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A C3 — TEST Lens
  Arms: TEST lens
Device: senofilcon A — CONTROL Lens
  Arms: CONTROL lens

SUMMARY:
This is a bilateral, dispensing, randomized, controlled, subject-masked, 2-arm parallel study to evaluate safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 39 (inclusive) years of age at the time of screening.
  4. By self-report, habitually wear spherical silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
  5. Have a habitual contact lens prescription that is current within the prior 6 months, and they must have worn that prescription for at least 2 weeks prior to entering the study.
  6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 through -6.00 D in both eyes.
  7. The subject's refractive cylinder must be 1.00 D or less.
  8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Have any ocular or systemic allergies or diseases that may interfere with contact lens wear.
  3. Have any autoimmune disease or use of medication, which may interfere with contact lens wear. Habitual medications used by successful soft contact lens wearers are considered acceptable.
  4. Have any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  5. Be currently wearing lenses in a monovision, multifocal, toric, or extended wear modality.
  6. Have participated in a contact lens or lens care product clinical trial within 14 days prior to study enrollment
  7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
  8. Have a history of binocular vision abnormality or strabismus.
  9. Have any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report. 10. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

  11. Have any ocular infection. 12. Have any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.

  13. Have entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (17):
- United States (17):
  - James T. Fujimoto, O.D., Cupertino, California
  - Randall Go, OD, San Francisco, California
  - Dr. James Weber & Associates, PA, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Flora Chen Poveda, OD, PA, Orange Park, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - VisualEyes, Inc, Roswell, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield Township, Michigan
  - Dr. Debbie H. Kim, OD, Closter, New Jersey
  - Sacco Eye Group, Vestal, New York
  - Professional Vision Care, Inc., Westerville, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Primary Eyecare Group, Brentwood, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - William J. Bogus, OD, FAAO, Salt Lake City, Utah
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 296 subjects were enrolled in this study. Of those enrolled, 295 subjects were dispensed at least one study lens, while 1 subject failed to meet all eligibility criteria. Of those dispensed, 289 subjects completed the study while 6 subjects were discontinued.
Groups:
- Control (Senofilcon A): Subjects that wore the Control (senofilcon A) lens during the study.
- Test (Senofilcon A C3): Subjects that wore the Test lens during the study.
Period: Overall Study
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Started | 150 | 145
Completed | 145 | 144
Not Completed | 5 | 1
Not completed — Subject enrolled in error | 1 | 0
Not completed — Study Procedure | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Subject no longer meets eligibility criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3) | Total
Number analyzed (Participants) | 150 | 145 | 295
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 30.0 (5.86) | 29.0 (5.70) | 29.5 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 102 | 100 | 202
  Gender: Male | 48 | 45 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 12 | 22
  Black or African American | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 131 | 122 | 253
  Multiple | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 150 | 145 | 295

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Vision Score
Description: Overall quality of vision score was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 145 | 144
Units on a scale | 67.0 (20.02) | 70.4 (19.73)
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculation using a two independent sample t test with a 2-sided type I error of 0.05, there would be enough power (i.e., 80%) for testing non-inferiority of the Test relative to the Control with 286 subjects (143 for each lens group) competing the study assuming the Test was 2 points higher than the Control; Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 2-sided 95% confidence interval of the mean difference was above -5; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = 3.1, 95% CI 2-sided [-0.6 to 6.7], Standard Error of Mean 1.86 — Least-square Mean difference was calculated as Test minus Control

2. Primary Outcome: Distance Monocular logMAR Visual Acuity
Description: Monocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale and was evaluated at distance (4 meter) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 145 | 144
Number analyzed (eyes) | 290 | 288
logMAR | -0.12 (0.093) | -0.11 (0.080)
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculation using a linear mixed model-based method with a 2-sided type I error of 0.05, there would be enough power (i.e., at least 80%) for testing non-inferiority of the Test relative to the Control with 16 subjects (8 for each lens group) competing the study assuming no difference between the Test and the Control; Test type: Non-Inferiority — Non-inferiority was declared if the upper bound of the 2-sided 95% confidence interval of the mean difference was below 0.05; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = 0.008, 95% CI 2-sided [-0.02 to 0.01], Standard Error of Mean 0.008 — Least-square Mean difference was calculated as Test minus Control

3. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits, 2-week follow-up and final evaluation). The data was then dichotomized into two groups. Those with Grade 3 or higher SLF and those with Grade 2 or lower. The proportion of eyes with Grade 3 or higher SLF was reported.
Time Frame: up to 2-week follow-up
Population: All subjects were dispensed at least one study lens. Subjects were summarized by actual treatment received.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 150 | 145
Number analyzed (eyes) | 300 | 290
proportion of eyes | 0 | 0
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculation using a simulation approach and Bayesian analysis with the 95% central posterior credible interval, there would be enough power (i.e., at least 80%) for assessing non-inferiority of the Test relative to the Control with 240 subjects (120 for each lens group) competing the study assuming no difference between the Test and the Control; Test type: Non-Inferiority — Non-inferiority was declared if the upper bound of the 95% central posterior credible interval of proportion difference was below 0.05; Bayesian hierarchical model; Mean Proportion Difference = 0.000, 95% CI 2-sided [-0.004 to 0.004], Standard Deviation 0.002 — Proportion difference was calculated as Test minus Control

4. Primary Outcome: Proportion of Eyes With Unacceptable Lens Fitting
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope post lens insertion and the 2-week follow-up. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The proportion of eyes with unacceptable lens fit was reported. Summaries presented in the Participant flow are summarized by planned arm, where as summaries for this measure are summarized by actual arm. One subject was dispensed the incorrect study lens, there for, the number of subjects that were randomized to the Control were 149 but 150 subjects were actually dispensed the control.
Time Frame: Up to 2-Week Follow-up
Population: All subjects were dispensed at least one study lens. Subjects were summarized by actual treatment received.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 150 | 145
Number analyzed (eyes) | 300 | 290
proportion of eyes | 0 | 0
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculation using a simulation approach and Bayesian analysis with the 95% central posterior credible interval, there would be enough power (i.e., at least 80%) for assessing non-inferiority of the Test relative to the Control with 140 subjects (70 for each lens group) competing the study assuming no difference between the Test and the Control; Test type: Non-Inferiority — Non- inferiority was declared if the upper bound of the 95% central posterior credible interval of proportion difference was below 0.1; Bayesian hierarchical model; Mean Proportion Difference = 0.000, 95% CI 2-sided [-0.004 to 0.004], Standard Deviation 0.002 — Proportion difference was calculated as Test minus Control

5. Secondary Outcome: Overall Comfort Scores
Description: Overall comfort scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 145 | 144
Units on a scale | 70.5 (22.83) | 70.4 (22.66)
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculated for the primary endpoints (i.e., 286 subjects with 143 per lens group), assuming the Test was 2 points higher than the Control, the estimated statistical power for testing non-inferiority of the Test relative to the Control was 73% for CLUE comfort using a two independent sample t test with a 2-sided type I error of 0.05; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -0.1, 95% CI 2-sided [-4.8 to 4.5], Standard Error of Mean 2.35 — Least-square Mean difference was calculated as Test minus Control

6. Secondary Outcome: Overall Handling Scores
Description: Overall handling scores were assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE handling score for each lens type was reported.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 145 | 144
Units on a scale | 69.2 (20.13) | 67.8 (20.44)
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculated for the primary endpoints (i.e., 286 subjects with 143 per lens group), assuming the Test was 2 points lower than the Control, the estimated statistical power for testing non-inferiority of the Test relative to the Control was 23% for CLUE handling using a two independent sample t test with a 2-sided type I error of 0.05; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Least-square Mean Difference = -1.9, 95% CI 2-sided [-6.0 to 2.3], Standard Error of Mean 2.13 — Least-square Mean difference was calculated as Test minus Control

7. Secondary Outcome: Situational Visual Performance - Indoors
Description: Indoor performance was assessed using the individual questionnaire item "Clarity of Vision indoors in bright light" with a 5-point Likert scale (1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor) and a Not Applicable response option. Subject responses were reported by lens using frequencies.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: number of responses
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 145 | 144
number of responses
  Not Applicable | 0 | 0
  Excellent | 75 | 85
  Very Good | 51 | 48
  Good | 17 | 11
  Fair | 1 | 0
  Poor | 1 | 0
Statistical Analysis 1: Comparison: Control (Senofilcon A) vs Test (Senofilcon A C3); Based on the sample size calculated for the primary endpoints (i.e., 286 subjects with 143 per lens group), assuming the percentage of "Excellent" rating for the Test was 10% higher than the Control, the estimated statistical power for testing non-inferiority of the Test relative to the Control was 93% using a Pearson chi-square test for two proportions with a 2-sided type I error of 0.05; Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the 2-sided 95% confidence interval of the odds ratio was greater than 0.67; Linear Mixed Model; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.83 to 2.16] — Odds Ratio was calculated as Test over Control

8. Secondary Outcome: Situational Visual Performance - Digital Devices
Description: Situational visual performance related to digital device use was assessed using the individual preference item "Overall preference while using computer screens & digital devices". The response set include: Strongly prefer my habitual lenses, Slightly prefer my habitual lenses, No Preference, Slightly prefer the study lenses and Strongly prefer the study lenses. Responses were collapsed into three categories for analysis purpose: Prefer Study Lens, No Preference, Prefer Habitual Lens. Subject responses were reported by lens using frequencies.
Time Frame: 2-Week Follow-up
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: number of responses
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
Number analyzed (Participants) | 146 | 144
number of responses
  Strongly prefer my habitual lenses | 17 | 12
  Slightly prefer my habitual lenses | 16 | 16
  No Preference | 61 | 48
  Slightly prefer the study lenses | 36 | 42
  Strongly prefer the study lenses | 16 | 26
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); Based on the sample size calculated for the primary endpoints (i.e., 286 subjects with 143 per lens group), assuming the percentage of subjects preferring Study lens was 20% higher than preferring Habitual lens in the Test lens group, the estimated statistical power for testing superiority of the Test relative to the Habitual was 88% using a simulation approach with a 2-sided type I error of 0.05; Test type: Superiority — Superiority was declared if the lower bound of the 2-sided 95% confidence interval of the preference ratio was greater than 1; Linear Mixed Model; Preference Ratio = 2.40, 95% CI 2-sided [1.40 to 4.10] — Preference ratio was calculated as Study lens over Habitual lens within the Test lens group

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 2 weeks.
Groups:
- Test (Senofilcon A C3): Subjects that wore the Test (senofilcon A C3) lens during the study.
Arm/Group | Control (Senofilcon A) | Test (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/145
Other Adverse Events (participants affected / at risk) | 0/150 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT05099380/Prot_SAP_000.pdf